CLINICAL TRIAL: NCT01446328
Title: Bergen Psychosis Project 2 - The Bergen-Stavanger-Innsbruck-Trondheim Study
Brief Title: Bergen Psychosis Project 2 - The Best Intro Study
Acronym: BP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Vest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/3387; 11/01070 (Other: The Norwegian Medicines Agency); 2010-022307-22 (EudraCT Number)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Antipsychotic Drugs; Randomized Controlled Trial; Treatment Effectiveness; Translational Research
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Amisulpride; Aripiprazole; Olanzapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amisulpride (Active Comparator)
  Interventions: Drug: Amisulpride
- Aripiprazole (Active Comparator)
  Interventions: Drug: Aripiprazole
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Amisulpride — Tablets, dose range 50-1200 mg/ day
  Other Names: Solian
  Arms: Amisulpride
Drug: Aripiprazole — Tablets, dose range 5-30 mg/ day
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Olanzapine — Tablets, dose range 2.5-20 mg/ day
  Other Names: Zyprexa
  Arms: Olanzapine

SUMMARY:
In the Bergen Psychosis Project 2 the antipsychotic drugs aripiprazole, amisulpride, and olanzapine will be compared head-to-head in patients with schizophrenia and related psychoses and followed for 12 months. The study is independent of the pharmaceutical industry, and in accordance with a pragmatic design a clinically relevant sample will be included with as few exclusion criteria as possible. The patients will be assessed repeatedly with regards to symptoms, side effects, and cognitive functioning, as well as laboratory parameters. The study hypothesis is that clinically meaningful differences among the drugs will be disclosed in a pragmatic design.

ELIGIBILITY:
Inclusion Criteria:

A:The observational cohort

* Patients 16 years old or older
* Active psychosis as determined by a score of 4 or more on one or more of the items Delusions, Hallucinatory behavior, Grandiosity, Suspiciousness/ persecution, or Unusual thought content in the Positive and Negative Syndrome Scale (PANSS).
* Or ICD-10 diagnosis corresponding to psychotic disorders or other mental disorders with psychotic features (F10-F19: .5 (psychotic disorder); F20-F29, F30.2, F31.2, F31.5, F32.3, F33.3). From which eligible patients are recruited to the B:The pragmatic, randomized, controlled trial (The Best Intro Study)
* Patients 18 years and older
* Schizophrenia spectrum and delusional disorder
* Symptoms of psychosis as determined by a score of 4 or more on one or more of the items Delusions, Hallucinatory behavior, Grandiosity, Suspiciousness/ persecution, or Unusual thought content in the Positive and Negative Syndrome Scale (PANSS).

Exclusion Criteria:

* Inability to understand spoken Norwegian.
* Patients with organic psychosis due to limbic encephalitis detected by antibodies in serum obtains at inclusion (such as NMDAR, VGKC and paraneoplastic antibodies performed at the Neuroimmunology Laboratory, Department of Neurology, Haukeland University Hospital) Pregnant or breast feeding women.
* Aripiprazole: Hypersensitivity to the active substance or to any of the excipients
* Amisulpride: Hypersensitivity to the active ingredient or to other ingredients of the medicinal product; concomitant prolactin-dependent tumours e.g. pituitary gland prolactinomas and breast cancer; phaeochromocytoma; lactation, combination with the following medications which could induce torsade de pointes: Class Ia antiarrhythmic agents such as quinidine, disopyramide, procainamide. Class III antiarrhythmic agents such as amiodarone, sotalol. Other medications such as bepridil, cisapride, sultopride, thioridazine, methadone, IV erythromycin, IV vincamine, halofantrine, pentamidine, sparfloxacin. Combinations with levodopa.
* Olanzapine: Hypersensitivity to the active substance or to any of the excipients. Patients with known risk of narrow-angle glaucoma.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change of the Positive and Negative Syndrome Scale total score | 12 months

SECONDARY OUTCOMES:
Change of the positive subscale scores of the Positive and Negative Syndrome Scale | 12 months
Change of the negative subscale scores of the Positive and Negative Syndrome Scale | 12 months
Change of the general subscale scores of the Positive and Negative Syndrome Scale | 12 months
Change of the Global Assessment of Functioning scale | 12 months
Change of the Clinical Global Impression - Severity of Illness score | 12 months
Change of the UKU Side Effects Rating Scale - Patient version score | 12 months
Change of serum High Density lipoprotein | 12 months
Change of serum Low Density lipoprotein | 12 months
Change of serum total cholesterols | 12 months
Change of serum triglycerides | 12 months
Change of serum fasting glucose | 12 months
Change of prolactin | 12 months
Change of the rate-corrected QT interval at electrocardiogram | 12 months
Change of body mass index | 12 months
  body weight in kilograms divided by the squared height in metres
Change of waist circumference | 12 months
Change of hip circumference | 12 months
Change of systolic blood pressure | 12 months
Change of diastolic blood pressure | 12 months

OTHER OUTCOMES:
Change of cognitive functions | 12 months
Change of mood symptoms | 12 months
Change of brain functional measures | 12 months
  Based on functional MRI - explorative
Change of brain structural measures | 12 months
  Based on structural MRI - explorative
Change of inflammatory markers in blood | 12 months
Change of gene expression in blood | 12 months
Change of bone turnover markers in serum | 12 months
Change of motor activity | 12 months
  Measured by actigraph
Change of autonomic activity | 12 months
  Measured by actiheart

CONTACTS AND LOCATIONS:
Overall Officials: Erik Johnsen, M.D., Ph.D., Principal Investigator — Haukeland University Hospital
Locations (4):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - St. Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Stabell LA, Johnsen E, Kroken RA, Loberg EM, Blindheim A, Joa I, Reitan SK, Rettenbacher M, Munk-Jorgensen P, Gjestad R. Clinical insight among persons with schizophrenia spectrum disorders treated with amisulpride, aripiprazole or olanzapine: a semi-randomised trial. BMC Psychiatry. 2023 Jun 29;23(1):482. doi: 10.1186/s12888-023-04981-9. PMID 37386462
- [Derived] Fathian F, Gjestad R, Kroken RA, Loberg EM, Reitan SK, Fleichhacker WW, Rettenbacher M, Larsen TK, Joa I, Stabell LA, Kjelby E, Sinkevicute I, Alisauskiene R, Steen VM, Johnsen E. Association between C-reactive protein levels and antipsychotic treatment during 12 months follow-up period after acute psychosis. Schizophr Res. 2022 Mar;241:174-183. doi: 10.1016/j.schres.2022.01.049. Epub 2022 Feb 4. PMID 35131596
- [Derived] Hoekstra S, Bartz-Johannessen C, Sinkeviciute I, Reitan SK, Kroken RA, Loberg EM, Larsen TK, Rettenbacher M, Johnsen E, Sommer IE. Sex differences in antipsychotic efficacy and side effects in schizophrenia spectrum disorder: results from the BeSt InTro study. NPJ Schizophr. 2021 Aug 18;7(1):39. doi: 10.1038/s41537-021-00170-3. PMID 34408155
- [Derived] Johnsen E, Kroken RA, Loberg EM, Rettenbacher M, Joa I, Larsen TK, Reitan SK, Walla B, Alisauskiene R, Anda LG, Bartz-Johannessen C, Berle JO, Bjarke J, Fathian F, Hugdahl K, Kjelby E, Sinkeviciute I, Skrede S, Stabell L, Steen VM, Fleischhacker WW. Amisulpride, aripiprazole, and olanzapine in patients with schizophrenia-spectrum disorders (BeSt InTro): a pragmatic, rater-blind, semi-randomised trial. Lancet Psychiatry. 2020 Nov;7(11):945-954. doi: 10.1016/S2215-0366(20)30341-2. PMID 33069317